CLINICAL TRIAL: NCT04250038
Title: Association of Cefepime Trough Levels With Clinical Efficacy and Neurotoxicity in Patients With Febrile Neutropenia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Matthias Gijsen, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62297
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Pharmacokinetics; Pharmacodynamics; Cefepime
Keywords: Cefepime; Pharmacokinetic; Neurotoxicity; Febrile neutropenia; Exposure
MeSH Terms: conditions — Neurotoxicity Syndromes; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective monocenter observational study, the objective was to determine a safe and effective therapeutic window for cefepime in patients with neutropenic fever.

DETAILED DESCRIPTION:
Cefepime, a fourth-generation cephalosporin, is widely prescribed for the treatment of serious bacterial infections. Cefepime has a more narrow spectrum and has relatively lower minimal inhibitory concentration (MIC) values compared to meropenem. Therefore cefepime is widely endorsed, and preferred over a carbapenem antibiotic, as a first line agent for the management of febrile neutropenia (FN) in hematologic patients.

Several studies have shown adequate exposure using the recommended 3x2 g dosing strategy for cefepime in most FN patients. The pharmacokinetic/pharmacodynamic (PKPD) target of fT100%>MIC, which is frequently used for BL AB in critically ill patients, is achieved in most patients. Subsets of patients have been shown to be at risk for underdosing, especially those with a higher than normal creatinine clearance, obese or cachectic patients and those infected with bacteria with a MIC >4 mg/L. Despite adequate cefepime exposure, the association with clinical outcome still needs to be confirmed on a large scale. An association between suboptimal PKPD target attainment and clinical outcome was shown on a large scale for β-lactam antibiotics. These data need to be validated for the specific antimicrobials agents and in subsets of patients. Another study suggested a cefepime PKPD target for clinical outcome of at least fT>MIC of 68% to 74% based on simulations using 2 existing population PK models. In a mixed population of critically and non-critically ill patients with Gram negative blood stream infections this threshold was a significant predictor of in-hospital mortality. A recent study, undertaken in patients with nosocomial pneumonia treated with cefepime, even reported clinical failure despite achievement of fT100%>MIC, they suggest a fCmin/MIC ratio of at least 2.1 as a better predictor for clinical failure in Gram negative bacterial pneumonia patients. Up until today, there are no explicit data linking PKPD target attainment with clinical outcome in FN patients.

With respect to cefepime toxicity, there is a lot of controversy on the upper limit that should not be exceeded in clinical practice. Cefepime toxicity is mainly neurological, going from mild confusion to seizures or encephalopathy. In the first study that assessed the relationship between cefepime PK and associated neurotoxicity, trough levels >22 mg/L were found to be associated with a 50% probability of neurological toxicity. However, a more recent study showed, using a non-parametric approach, that estimated rates of neurotoxicity using this threshold are very high and discordant with rates seen in clinical practice. Hence this threshold seems not representative for the clinical practice. Other PK parameters (Cmax, AUC, ...) and covariates (CrCl, Age, dose, duration of therapy, co-medication, …) probably also influence cefepime related neurotoxicity. Recently, an attempt to redefine cefepime's threshold for neurotoxicity was published in a retrospective cohort study. No neurotoxicity was observed below 35 mg/L for all samples (steady-state levels during continuous infusion, trough and non-trough levels during intermittent infusion). However, when looking only at trough levels, they also advise avoiding levels >20 mg/L until more information from prospective studies is available.

Moreover, until now there has only been one study investigating the carryover of cefepime in samples taken via a central venous catheter. This study suggested possible carryover for triple lumen catheters and peripherally-inserted central catheters. Due to the small sample size and the in vitro nature of this research, these results need to be confirmed.

The aim of this research is two-fold. Firstly, the aim is to investigate whether there is significant carryover of cefepime in samples taken via a central venous catheter. Next, the aim is to assess prospectively the relation between cefepime exposure and efficacy or safety in a FN patient population. As literature on these topics is scarce this research will further explore the exposure-response relationship in order to define a therapeutic window for maximal clinical cure and minimal neurotoxicity that can be used in future research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the hemato-oncology ward
* treated with cefepime for neutropenic fever
* written informed consent

Exclusion Criteria:

- younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemato-oncology patients treated with cefepime for neutropenic fever
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic failure | From Day 2 before until Day 2 day after day of sampling
  hemoculture positive for Gram negative bacteria during cefepime therapy
Neurotoxicity: cognitive disturbance, confusion, depressed level of consciousness, encephalopathy, hallucinations, movements involuntary, seizure | From Day 2 before until Day 2 day after day of sampling
  Percent of patients and trough levels associated with one of following symptoms during cefepime therapy: cognitive disturbance, confusion, depressed level of consciousness, encephalopathy, hallucinations, movements involuntary, seizure
Carryover cefepime in samples via central venous catheter | From Day 2 before until Day 2 day after day of sampling
  Difference between cefepime concentration in samples obtained via central venous catheter vs. samples obtained via peripheral venipuncture

SECONDARY OUTCOMES:
Fever | From Day 2 before until Day 2 day after day of sampling
  Presence of fever per day of treatment, defined as T° above 38°C on two occasions (min. 1h apart) or above 38.3°C on one occasion
Clinical condition | From Day 2 before until Day 2 day after day of sampling
  Evolution in clinical condition compared to the previous day as evaluated by the treating physician, per day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Study Director — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be discussed upon reasonable request

REFERENCES:
- [Background] Roberts JA, Paul SK, Akova M, Bassetti M, De Waele JJ, Dimopoulos G, Kaukonen KM, Koulenti D, Martin C, Montravers P, Rello J, Rhodes A, Starr T, Wallis SC, Lipman J; DALI Study. DALI: defining antibiotic levels in intensive care unit patients: are current beta-lactam antibiotic doses sufficient for critically ill patients? Clin Infect Dis. 2014 Apr;58(8):1072-83. doi: 10.1093/cid/ciu027. Epub 2014 Jan 14. PMID 24429437
- [Background] Rhodes NJ, Kuti JL, Nicolau DP, Van Wart S, Nicasio AM, Liu J, Lee BJ, Neely MN, Scheetz MH. Defining Clinical Exposures of Cefepime for Gram-Negative Bloodstream Infections That Are Associated with Improved Survival. Antimicrob Agents Chemother. 2015 Dec 14;60(3):1401-10. doi: 10.1128/AAC.01956-15. PMID 26666929
- [Background] Aitken SL, Altshuler J, Guervil DJ, Hirsch EB, Ostrosky-Zeichner LL, Ericsson CD, Tam VH. Cefepime free minimum concentration to minimum inhibitory concentration (fCmin/MIC) ratio predicts clinical failure in patients with Gram-negative bacterial pneumonia. Int J Antimicrob Agents. 2015 May;45(5):541-4. doi: 10.1016/j.ijantimicag.2014.12.018. Epub 2015 Jan 19. PMID 25665726
- [Background] Lamoth F, Buclin T, Pascual A, Vora S, Bolay S, Decosterd LA, Calandra T, Marchetti O. High cefepime plasma concentrations and neurological toxicity in febrile neutropenic patients with mild impairment of renal function. Antimicrob Agents Chemother. 2010 Oct;54(10):4360-7. doi: 10.1128/AAC.01595-08. Epub 2010 Jul 12. PMID 20625153
- [Background] Rhodes NJ, Kuti JL, Nicolau DP, Neely MN, Nicasio AM, Scheetz MH. An exploratory analysis of the ability of a cefepime trough concentration greater than 22 mg/L to predict neurotoxicity. J Infect Chemother. 2016 Feb;22(2):78-83. doi: 10.1016/j.jiac.2015.10.009. Epub 2015 Dec 17. PMID 26712584
- [Background] Huwyler T, Lenggenhager L, Abbas M, Ing Lorenzini K, Hughes S, Huttner B, Karmime A, Uckay I, von Dach E, Lescuyer P, Harbarth S, Huttner A. Cefepime plasma concentrations and clinical toxicity: a retrospective cohort study. Clin Microbiol Infect. 2017 Jul;23(7):454-459. doi: 10.1016/j.cmi.2017.01.005. Epub 2017 Jan 19. PMID 28111294
- [Background] Marsh E, Verhoven SM, Groszek JJ, Fissell WH, An G, Patel P, Creech B, Shotwell M. Beta-lactam carryover in arterial and central venous catheters is negligible. Clin Chim Acta. 2018 Nov;486:265-268. doi: 10.1016/j.cca.2018.08.008. Epub 2018 Aug 15. PMID 30118674